CLINICAL TRIAL: NCT00962013
Title: A Prospective Open-Label Evaluation of the Restoration® Modular System
Brief Title: Restoration® Modular Revision Hip System Post Market Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53
Record Dates: First submitted 2009-08-13; First posted 2009-08-19 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restoration® Modular (Other): All subjects were enrolled into a single arm and received the Restoration® Modular Revision Hip System to replace the femoral portion of a failed previous implant.
  Interventions: Device: Restoration® Modular Revision Hip System

INTERVENTIONS:
Device: Restoration® Modular Revision Hip System — Restoration® Modular Revision System

SUMMARY:
The purpose of this study is to demonstrate survivorship of the femoral stem at 5 years.

DETAILED DESCRIPTION:
The two-piece modular revision stem components are intended to be used for primary or revision total hip arthroplasty, as well as in the presence of severe proximal bone loss. This study evaluates the System in revision cases only. The stems are intended to be used with Stryker Orthopaedics femoral heads, unipolar and bipolar components, and acetabular components. These femoral stems are designed to be press fit into the proximal femur.

In addition to demonstrating survivorship at 5 years, this study will seek to gain information on four secondary objectives: radiographic stability, Harris Hip Scores, SF-36 general well-being assessment, and safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for cementless revision of a failed femoral prosthesis.
* Patients willing to sign the informed consent.
* Patients able to comply with follow-up requirements including post-operative weightbearing restrictions and self-evaluations.
* Male and non-pregnant female patients ages 18 to 85 years of age at the time of surgery.

Exclusion Criteria:

* Patients with ongoing infection.
* Patients who are severely immunocompromised.
* Patients who are prisoners.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2004-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Barnett, MD, Principal Investigator — Orthopaedic Specialty Institute; Michael W Britt, MD, Principal Investigator — Orthopaedic Associates of Corpus Christi; Kenneth A Greene, MD, Principal Investigator — Crystal Clinic; Steven F Harwin, MD, Principal Investigator — Beth Israel Medical Center; D. Christopher Hikes, MD, Principal Investigator — Providence Health & Services; Kirby Hitt, MD, Principal Investigator — Scott and White Hospital; William Hozack, md, Principal Investigator — Rothman Institute; Frederick Jaffe, MD, Principal Investigator — Hospital for Joint Diseases; Timothy P Lovell, MD, Principal Investigator — Providence Orthopaedic Specialties; Mark R Matthes, MD, Principal Investigator — Iowa Orthopaedic Center; Arthur Malkani, MD, Principal Investigator — Jewish Hospital Center for Advanced Medicine; John Schurman, MD, Principal Investigator — Kansas Joint and Spine Institute; John Wright, MD, Principal Investigator — New West Sports Medicine and Orthopaedic Surgery
Locations (13):
- United States (13):
  - Orthopaedic Specialty Institute, Orange, California
  - Iowa Orthopaedic Center, Des Moines, Iowa
  - Kansas Joint and Spine Institute, Wichita, Kansas
  - Jewish Hospital Center for Advanced Medicine, Louisville, Kentucky
  - New West Sports Medicine and Orthopaedic Surgery, Kearney, Nebraska
  - Hospital for Joint Diseases, New York, New York
  - Beth Israel Medical Center, New York, New York
  - Crystal Clinic, Akron, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Rothman Institute, Philadelphia, Pennsylvania
  - Orthopedic Associates of Corpus Christi, Corpus Christi, Texas
  - Scott and White Hospital, Temple, Texas
  - Providence Orthopaedic Specialities, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 137/139 participants/hips enrolled and 17/17 participants/hips censored=120/122 participants/hips started
Period: Overall Study
Arm/Group | Restoration® Modular
Started | 120
Completed | 52 (Number of participants with 5 year primary endpoint data)
Not Completed | 68
Not completed — Did not have surgery | 1
Not completed — Death | 8
Not completed — Lost to Follow-up | 12
Not completed — Unable/Unwilling to return | 6
Not completed — Withdrawal by Subject | 8
Not completed — Removal of study device | 3
Not completed — Site Termination | 24
Not completed — No 5 year evaluation | 6

BASELINE CHARACTERISTICS:
Population: Includes participants who received the Restoration® Modular Hip System and were not censored from analysis.
Arm/Group | Restoration® Modular
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] — Age results are based on 118 participants as there were 2 participants missing age data. For bilateral participants, age at the time surgery for the first hip enrolled is used for the baseline measurement.
  years | 67.72 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 59
Region of Enrollment [Number; unit: participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: Stem Survivorship (%)
Description: Failure is defined by stem revision for any cause.
Time Frame: 5 years
Population: Participants with 5 year follow-up evaluations or participant had a stem revision before they reached 5 years.
Measure: Number (90% Confidence Interval); unit: stem survivorship percentage at 5 years
Units Other Than Participants: hips
Groups:
- Restoration® Modular: All subjects were enrolled into a single arm and received the Restoration Modular Revision Hip System to replace the femoral portion of a failed previous implant.
Arm/Group | Restoration® Modular
Number analyzed (Participants) | 55
Number analyzed (hips) | 56
stem survivorship percentage at 5 years | 94.64 [89.69 to 99.59]
Statistical Analysis 1: Comparison: Restoration® Modular; This revision study will demonstrate a 5-year survivorship of the Restoration Modular system not seven percent worse than an expected 95% survival rate using a lower 95% one-sided confidence bound; Test type: Non-Inferiority or Equivalence — non-inferiority margin is 7%; p = 0.0136, Exact Binomial

2. Secondary Outcome: Radiographic Stability
Description: Absence of a radiolucent lines ≥ 2mm around the entire stem in AP or ML view.
Time Frame: 5 years
Population: 41 hips had fully evaluable radiographs at the 5 year interval; 40 out of the 41 hips are stable.
Measure: Number (95% Confidence Interval); unit: percentage of stable hips
Units Other Than Participants: hips
Arm/Group | Restoration® Modular
Number analyzed (Participants) | 40
Number analyzed (hips) | 41
percentage of stable hips | 97.6 [87.1 to 99.9]

3. Secondary Outcome: Harris Hip Score
Description: Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score less than or equal to 79 is considered fair-poor.
  90 - 100 = excellent
  80 - 89 = good
  70 - 79 = fair
  0 - 69 = poor
Time Frame: pre-op and 5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | Restoration® Modular
Number analyzed (Participants) | 110
Number analyzed (hips) | 110
units on a scale
  Mean HHS Pre-op N=110 | 46.33 (16.34)
  Mean HHS 5 years N=45 | 88.27 (10.91)
Statistical Analysis 1: Comparison: Restoration® Modular; Change from HHS pre-op to HHS 5 year; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: SF-36 Health Status Survey: Role - Physical
Description: Consists of 8 subscores all with a range of 0-100; a higher score indicates a better health state:
  The subscores are: 1 - Physical Functioning, 2 - Role-Physical, 3 - Bodily Pain, 4 - General Health, 5 - Vitality, 6 - Social Functioning, 7- Role-Emotional, 8 - Mental Health
  This Secondary Outcome Measure is focused on the "Role-Physical" score.
Time Frame: pre-op, 2 year and 5 year
Population: SF-36 Scores were assessed for each hip. (One hip did not have a pre-operative SF-36)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | Restoration® Modular
Number analyzed (Participants) | 120
Number analyzed (hips) | 121
units on a scale
  SF-36 Role-Physical Pre-op N=121 | 31.21 (10.67)
  SF-36 Role-Physical 2 year N=86 | 42.25 (12.15)
  SF-36 Role-Physical 5 year N=45 | 44.66 (13.24)
Statistical Analysis 1: Comparison: Restoration® Modular; Change from SF-36 Role-Physical pre-op score to 2 and 5 year scores; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

5. Primary Outcome: Femoral Stem Fracture
Time Frame: 5 years
Population: Participants who received the Restoration Modular Hip System.
Measure: Number; unit: femoral stem fractures
Arm/Group | Restoration® Modular
Number analyzed (Participants) | 120
femoral stem fractures | 0

6. Secondary Outcome: Post-surgery Femoral Crack/Fracture and Subsidence Rate
Time Frame: Post-op to 5 years
Population: Post-surgery femoral crack/fracture and subsidence rate were assessed by hip.
Measure: Number; unit: percentage of hips
Units Other Than Participants: hips
Arm/Group | Restoration® Modular
Number analyzed (Participants) | 120
Number analyzed (hips) | 122
percentage of hips
  Post-surgery femoral stem crack/fracture rate % | 1.64
  Femoral subsidence rate % | 1.64
Statistical Analysis 1: Comparison: Restoration® Modular; Post-surgery femoral stem crack/fracture rate compared to 21% (pre-specified in protocol based on literature rates) Femoral subsidence rate compared to 18% (pre-specified in protocol based on literature rates); Test type: Superiority or Other; p < 0.0001, Exact Binomial

ADVERSE EVENTS:
Time Frame: Enrollment to 5 years post-op. Censored protocol violations not included as at risk participants. Industry standard Adverse Event (AE) terms (e.g. MedDRA) were not used for AE data collection. Specific AE terms were not used for all AEs collected.
Description: Serious AEs & AEs related to the implant/procedure collected. Elective procedures not included. i.e. non-study joint replacement/revision, rotator cuff repair, carpal tunnel release, cataract, intra-ocular & bunion procedures, total shoulder repair, laminectomy, microdiscectomy, breast reduction, cervical spine fusion, & mid-foot/flat-foot surgery.
Arm/Group | Restoration® Modular
Serious Adverse Events (participants affected / at risk) | 44/120
Other Adverse Events (participants affected / at risk) | 44/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restoration® Modular (N=120)
Non-operative Site Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 5 (7)
Non-operative Site Cardiac Disorders (Cardiac disorders) | 9 (16)
Non-operative Site Gastrointestinal Disorders (Gastrointestinal disorders) | 8 (11)
Non-operative Site General Disorders (General disorders) | 2 (2)
Non-operative Site Hepatobiliary Disorders (Hepatobiliary disorders) | 1 (1)
Non-operative Site Infections and Infestations (Infections and infestations) | 8 (11)
Operative Site Infections or Infestations (Infections and infestations) | 6 (8)
Non-operative Site Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 1 (2)
Operative Site Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 2 (2)
Non-operative Site Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 7 (9)
Operative Site Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 17 (22)
Non-Operative Site Neoplasms Benigh, Malignant, and Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Non-operative Site Nervous System Disorders (Nervous system disorders) | 4 (5)
Non-operative Site Renal and Urinary Disorders (Renal and urinary disorders) | 2 (2)
Non-operative Site Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Non-operative Site Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Non-operative Site Vascular Disorders (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restoration® Modular (N=120)
Operative Site Injury,Poisoning and Procedural Complication (Injury, poisoning and procedural complications) | 6 (7)
Non-operative Site Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 9 (10)
Operative Site Musculoskeleatal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 35 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results at the completion of the study.These manuscripts and abstracts will be delayed until after the multi-center publication is submitted.All publications shall be submitted to the Sponsor for review at least 60 days prior to submission of publication.The Sponsor shall not edit or otherwise influence the publications other than to ensure that confidential information is not disclosed and that the data is accurately represented.